CLINICAL TRIAL: NCT00311974
Title: The Effect of Dihydralazine on Renal Tubular Function and Vasoactive Hormones in Healthy Individuals
Brief Title: The Effect of Dihydralazine on Kidney Function and Hormones in Healthy Individuals
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Regional Hospital Holstebro (Other)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: MED.RES.HOS.2006.01.HV; 99127500
Record Dates: First submitted 2006-04-05; First posted 2006-04-07 (Estimated); Last update posted 2010-02-18 (Estimated); Status verified 2010-02

CONDITIONS: Healthy
Keywords: Dihydralazine; Sympathetic activation; Fractional sodium excretion
MeSH Terms: interventions — Dihydralazine

INTERVENTIONS:
Drug: Dihydralazine

SUMMARY:
We, the investigators at Holstebro Hospital, want to test the hypothesis that dihydralazine leads to the activation of the sympathetic nervous system in healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Men
2. Ages 18 to 40 years.
3. Body mass index less than or equal to 30 kg/m2

Exclusion Criteria:

1. History or clinical signs of heart, lung, kidney, or endocrine organ disease.
2. Abnormal biochemical screening of the blood regarding: B-hemoglobin, P-sodium, P-potassium, P-creatinine, P-albumin, P-bilirubin, P-alanine aminotransferase, P-alkaline phosphatase, P-cholesterol, and B-glucose.
3. Abnormal screening of the urine regarding: albumin and glucose
4. Malignant disease.
5. Known arterial hypertension or measured 24 hour blood pressure above 135 mmHg systolic or 85 mmHg diastolic.
6. Alcohol abuse.
7. Smoking.
8. Drug use or abuse.
9. Known intolerance or allergy to dihydralazine
10. Blood donation within 1 month of the start of the study.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16
Dates: Start 2006-04; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Fractional sodium excretion
Heart rate
Blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Erling B Pedersen, Professor, Study Chair — Department of Medical Research, Holstebro Hospital, Denmark; Henrik Vase, MD, Principal Investigator — Department of Medical Research, Holstebro Hospital, Denmark
Locations (1):
- Department of Medical Research, Holstebro Hospital, Holstebro, Denmark